CLINICAL TRIAL: NCT00507039
Title: Repeatability of a Single Concentration and Single-step Bronchial Allergen Challenge With Grass Pollen
Brief Title: Safety and Repeatability of Bronchial Challenge With Grass-pollen
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Johannes Schulze MD, Cosultant Pediatric Allergy and Pulmonology, Johann Wolfgang Goethe University Hospital
Other Study IDs: 334/06/FFM
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Allergic Asthma
Keywords: PD20 FEV1; grass pollen; one-step

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- grass allergy, bronchial challenge: subjects with known allergy against grass-pollen undergo bronchial challenges
  Interventions: Procedure: inhalative grass-pollen provocation

INTERVENTIONS:
Procedure: inhalative grass-pollen provocation — Subjects undergo allergen challenges with incremental doses of grass pollen allergen. In subjects, who develop a fall in FEV1 of more than 20%, this will be followed by two single-step challenges.
  Other Names: Viasys APS, Allergopharma allergen

SUMMARY:
The study is meant to establish a one-step challenge with grass-pollen in patients sensitized for grass-pollen. Therefore the investigators compare a multi-step challenge with grass-pollen with an one-step challenge in order to survey the repeatability and safety.

DETAILED DESCRIPTION:
Background:

Specific provocation with inhaled allergens is an established tool in clinical practice and research, supporting the understanding of pathophysiology of allergic asthma, and analysing the efficacy of new therapies. This study examines the repeatability of a bolus-dose inhalative allergen challenge with grass pollen.

Method:

Forty grass pollen allergics should undergo an incremental-dose grass pollen challenge to calculate their PD20-dose. This calculated dose will be applicated twice to analyse the repeatability of the bolus dose challenge. Before and twenty-four hours after the provocation, exhaled nitric oxid (FeNO) will be determined as a marker of bronchial inflammation.

ELIGIBILITY:
Inclusion Criteria:

* age >12 <45 years
* known sensitization for grass-pollen
* informed consent

Exclusion Criteria:

* age <12 >45 years
* clinical asthma requiring regular inhalation
* vital capacity <80%
* FEV1 < 75%
* chronic disease conditions or infections
* pregnancy
* inhalative or systemic steroid use
* substance abuse
* incapability of understanding the study's purpose and performance

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects undergo allergen challenges with incremental doses of grass pollen allergen. In those subjects, who develop a fall in FEV1 of more than 20%, this is followed by two single-step challenges in an interval of at least seven days.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2007-02; Primary Completion 2008-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
repeatability of a bolus-dose inhalative allergen challenge with grass pollen | feb 2007 - aug 2008

SECONDARY OUTCOMES:
kappa-index of concordance: reliability of the three procedures titrated skin prick-test, incremental challenge and bolus challenge with grass pollen. | feb 2007 - dec 2007

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, M.D., Ph.D, Principal Investigator — Goethe University, Department of Pulmonology
Locations (1):
- Goethe University, Department of Pulmonology, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Cockcroft DW, Ruffin RE, Frith PA, Cartier A, Juniper EF, Dolovich J, Hargreave FE. Determinants of allergen-induced asthma: dose of allergen, circulating IgE antibody concentration, and bronchial responsiveness to inhaled histamine. Am Rev Respir Dis. 1979 Nov;120(5):1053-8. doi: 10.1164/arrd.1979.120.5.1053. No abstract available. PMID 507521
- [Background] Cockcroft DW, Murdock KY, Kirby J, Hargreave F. Prediction of airway responsiveness to allergen from skin sensitivity to allergen and airway responsiveness to histamine. Am Rev Respir Dis. 1987 Jan;135(1):264-7. doi: 10.1164/arrd.1987.135.1.264. PMID 3800152